CLINICAL TRIAL: NCT02014818
Title: Multicenter Comparison of Early and Late Vascular Responses to Everolimus-eluting Cobalt-CHromium Stent and Platelet AggregatioN Studies In Patients With Stable Angina Managed as Elective Case : MECHANISM-Elective
Brief Title: Multicenter Comparison of Early and Late Vascular Responses to Everolimus-eluting Cobalt-CHromium Stent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kobe University (Industry)
Responsible Party: Principal Investigator, Toshiro Shinke, MD, PhD, Associate Professor, Kobe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MECHANISM-Elective
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This study will comprise of 1 month follow-up and 3-month follow up arm, which enroll patients in a parallel manner.
Who Masked: Outcomes Assessor
Masking Description: All patients' information will be blinded to OCT image analyzers.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3 month OCT follow-up, CoCr-EES (Experimental): Elective PCI can be performed with the use of an EES. PCI in another vessel or follow-up angiography is expected to be performed 3 months after the index procedure.
  Interventions: Device: CoCr-EES
- 1 month OCT follow-up, CoCr-EES (Experimental): Elective PCI can be performed with the use of an EES. PCI in another vessel or follow-up angiography is expected to be performed 1 months after the index procedure.
  Interventions: Device: CoCr-EES

INTERVENTIONS:
Device: CoCr-EES
  Other Names: XIENCE PRIME; XIENCE Xpedition

SUMMARY:
To treat patients with stable coronary artery disease, elective percutaneous coronary intervention (PCI) will be performed with the use of an everolimus-eluting cobalt- chromium stent (everolimus-eluting stent: EES, Xience Prime, Xpedition), which is the current standard drug-eluting stent (DES). Vascular responses at the site of stent placement will be evaluated by optical coherence tomography (OCT) at 1 or 3 months and at 12 months after stent placement, along with observation of changes over time in the target vessel. The relationships between OCT findings and the time course of platelet aggregation and between OCT findings and the occurrence of major cardio- cerebrovascular events will also be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Patients having at least one de novo lesion in a coronary artery in whom PCI with a DES is indicated
* Patients aged 20 to less than 85 years at the time of informed consent
* Patients who have provided informed consent written by themselves
* Patients who are able to undergo OCT examinations of the site of stent placement at 1 or 3 months and at 12 months

Exclusion Criteria:

* If it is judged difficult to perform clinical and angiographic follow-up at 12 months (considering the patient's remote place of residence, etc.)
* Patients with acute myocardial infarction (AMI)
* Patients in a state of shock
* Patients with cardiac failure
* Patients having a culprit lesion in the left main coronary artery trunk
* Patients having a lesion with a reference vessel diameter of less than 2.0 mm or 4.5 mm or larger by visual estimate
* Patients having an in-stent restenosis lesion as the culprit lesion
* Patients having chronic renal failure with a serum creatinine level of 2.0 mg/dL or higher at a screening visit
* Patients on hemodialysis
* Cancer patients with a life expectancy of less than 2 years
* Patients who are scheduled to undergo elective surgery requiring discontinuation of antiplatelet therapy within the next 3 months
* Pregnant women or women expected to become pregnant
* Patients with a history of adverse reactions to aspirin or clopidogrel (however, it is acceptable to enroll patients in whom the safety of ticlopidine has been confirmed, even if they have a history of adverse reactions to clopidogrel)

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of stent-strut coverage determined by OCT. | 3 months
  Rate of stent-strut coverage determined by OCT at 3 months after stent placement (To observe temporal course from the early stage, the rate of stent-strut coverage in the 1-month arm will also be evaluated in a complementary manner, separately from the 3-month arm.) To identify the factors defining the strut coverage at 1-month or 3-months, from OCT index, blood markers, platelet aggregation test immediately after stenting, the strut coverage of 1 to 3 months

SECONDARY OUTCOMES:
All-cause Death, Cardiac death, MI, Stroke, Major bleeding | 1-year
  All-cause Death, Cardiac death, MI, Stroke, Major bleeding
Any TLR | 1-year
  Any target lesion revascularization at 1-year
Clinically-driven TLR | 1 year
  Clinically relevant revascularization, such as ischemia driven intervention
Any TVR | 1 year
  Any target vessel revascularization including both target lesion and remote lesion.
CABG | 1 year
  Coronary artery bypass grafting
Any revascularization | 1 year
  Any revascularization including percutaneous intervention and surgical bypass grafting
Angiographic binary restenosis | 12 month
  Angiographic restenosis defined as percentage of diameter stenosis more than 50% at target lesion
Patient-oriented composite | 1 year
  All-cause death, Any MI including non-target territory, Any repeat revascularization
  ,Stroke
The percentage of stent strut coverage by OCT | 12 month
  Determination of factors associated with 12-month rate of stent-strut coverage on the basis of OCT findings, circulating biomarkers, and platelet aggregation test results immediately after stent placement
OCT endpoint | 1-month or 3-month
  * The percentage of stent strut malapposition
  * The presence of Intra-stent thrombus
  * Intra-stent thrombus area (Maximum site)
  * Intra-stent thrombus length
  * The number of Intra-stent thrombus
Angiographic Quantitative analysis | 12 month
  * In-segment late loss
  * Minimal lumen diameter (MLD), reference vessel diameter (RVD), percent diameter stenosis (%DS)
  * In-stent late loss
  * Binary restenosis (In-stent, In-segment, Peri-stent)
  * Angiographically detected stent fracture（based on Popma's classification ）
Angiographic Qualitative analysis | 12 month
  * Peri-stent contrast stain (PSS)
  * Site and pattern of restenosis (based on Mehran clasification)

OTHER OUTCOMES:
Platelet Aggregation Test | At the time of OCT follow-up (1 month or 3 month) and 12 month
  (1) at the time of PCI, (2) at the time of OCT at 1 or 3 months after PCI, (3) at 12-month follow-up, and (4) at the time of occurrence of a cardio-cerebrovascular event.

CONTACTS AND LOCATIONS:
Overall Officials: Toshiro Shinke, MD, PhD, Principal Investigator — Kobe University Graduate School of Medicine
Locations (1):
- Kobe University Graduate School of Medicine, Kobe, Japan